CLINICAL TRIAL: NCT05863156
Title: Evaluation of the Effects of Different Positions Given During Antenatal Electro-Fetal Monitoring on Maternal Comfort, Maternal Blood Pressure and Fetal Health
Brief Title: Evaluation of the Effects of Different Positions Given During Antenatal Electro-Fetal Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Tuğba YILMAZ ESENCAN, Vice-dean, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NST
Record Dates: First submitted 2023-03-28; First posted 2023-05-17 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Fetal Monitoring; Patient Comfort; Maternal Health
Keywords: Fetal Monitoring; Patient Comfort; Maternal Health; Midwifery

STUDY DESIGN:
Intervention Model Description: The study was conducted in a pregnant follow-up outpatient clinic of a maternity hospital in Istanbul, between December 2021 and January 2023, in a randomized controlled experimental study design with two interventions and a control group. In the study, 60 participants were placed in the right side lying position (intervention 1), 60 participants in the semi-sitting position (intervention 2) and 120 participants in the left side lying position (control group), and the study was completed with a total of 240 pregnant women. Research data were collected through the Information Form and the General Comfort Scale-Short Form.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention 1 (Experimental): electro fetal monitoring
  Interventions: Diagnostic Test: Right side lying position; Diagnostic Test: Semi Fowler; Diagnostic Test: left side lying position
- intervention 2 (Experimental): electro fetal monitoring
  Interventions: Diagnostic Test: Right side lying position; Diagnostic Test: Semi Fowler; Diagnostic Test: left side lying position
- control group (Experimental): electro fetal monitoring
  Interventions: Diagnostic Test: Right side lying position; Diagnostic Test: Semi Fowler; Diagnostic Test: left side lying position

INTERVENTIONS:
Diagnostic Test: Right side lying position — In the study, 60 participants were placed in the right side lying position (intervention 1)
  Other Names: (intervention 1)
Diagnostic Test: Semi Fowler — In the study, 60 participants in the semi-sitting position (intervention 2)
  Other Names: (intervention 2)
Diagnostic Test: left side lying position — In the study, 120 participants in the left side lying position (control group).
  Other Names: (control group)

SUMMARY:
The objective of this study was to assess the effects of different maternal positions during electronic fetal monitoring (EFM) on maternal and fetal health outcomes. The study was conducted between December 2021 and January 2023 in a maternity hospital in Istanbul, employing a randomized controlled trial design. A total of 240 pregnant women were randomized into three groups: 60 participants were assigned to the right-side lying position (intervention 1), 60 to the semi-sitting position (intervention 2), and 120 to the left-side lying.

Maternal systolic blood pressure, body temperature, and pulse rate were measured before, during, and after the EFM procedure. Research data were collected through the Information Form and the General Comfort Scale-Short Form.

DETAILED DESCRIPTION:
IIntroduction: Electronic fetal monitoring (EFM) is widely utilized for pregnancy and labor management due to its non-invasive nature, ease of use, and accessibility. However, the accuracy of EFM outcomes may be influenced by various factors, including the maternal position during monitoring, maternal comfort, and maternal blood pressure. This study aimed to explore how different positions during EFM influence both maternal.

Objective: The primary objective of this study was to examine the effects of three different maternal positions during EFM-right-side lying, semi-sitting, and left-side lying-on maternal and fetal health parameters. These parameters included systolic blood pressure, body temperature, pulse rate, and maternal comfort.

Methods:

A randomized controlled trial was conducted in a pregnancy follow-up outpatient clinic at a maternity hospital in Istanbul from December 2021 to January 2023. The study included 240 pregnant women, who were randomly assigned to one of three groups:

* Intervention 1 (right-side lying position) - 60 participants
* Intervention 2 (semi-sitting position) - 60 participants
* Control group (left-side lying position) - 120 participants Maternal physiological data were collected at three time points: pre-EFM, during EFM, and post-EFM. The General Comfort Scale-Short Form was used to assess maternal comfort. Statistical analyses were conducted to identify significant differences between groups and over time.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18,
* Being 35 years of age and under,
* Being a single fetus in the late 3rd trimester (34th-40th gestational week),
* Fetal biometric measurements between 34-40 weeks of gestation,
* No maternal and fetal risk affecting pregnancy,
* It was determined that the vital signs were within normal values before the application, not being hungry during the application (at the latest 2 hours of fasting time will be checked), and accepting the recommended application position.

Exclusion Criteria:

- The pregnant woman does not accept the recommended application position.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 305 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: TUĞBA YILMAZ ESENCAN, Principal Investigator — Uskudar University
Locations (1):
- Uskudar Univercity, Istanbul, Ümraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Humphries A, Mirjalili SA, Tarr GP, Thompson JMD, Stone P. The effect of supine positioning on maternal hemodynamics during late pregnancy. J Matern Fetal Neonatal Med. 2019 Dec;32(23):3923-3930. doi: 10.1080/14767058.2018.1478958. Epub 2018 Jun 3. PMID 29772936
- [Derived] Yilmaz Esencan T, Demir Yildirim A, Sagiroglu E. Effects of maternal positions in electronic fetal monitoring: a randomised controlled trial. BMC Nurs. 2025 Jan 7;24(1):22. doi: 10.1186/s12912-024-02654-w. PMID 39773730

RESULTS

PARTICIPANT FLOW:
Recruitment Details: December 2021 - January 2023
Pre-assignment Details: Randomization for the study was carried out on the website random.org; unique values were generated to divide 305 into 2 unique groups. The first group of 161 (81+81) numbers was randomly assigned to the intervention group, while the second group of 143 numbers was assigned to the control group.
Groups:
- The Right Lateral Position; The Semi-Fowler Position; Control Group: the Left Lateral Position: electro fetal monitoring
  Right side lying position: In the study, 60 participants were placed in the right side lying position (intervention 1)
  Semi Fowler: In the study, 60 participants in the semi-sitting position (intervention 2)
  left side lying position: In the study, 120 participants in the left side lying position (control group).
Period: Overall Study
Arm/Group | The Right Lateral Position | The Semi-Fowler Position | Control Group: the Left Lateral Position
Started | 81 (The intervention group, which was fixed at 120 pregnant woman, was divided into two subgroups in which 60 women were placed in the right lateral side-lying position (Intervention 1) Allocated to intervention (n=81): Received allocated intervention (n=60) It was excluded because of insufficient follow-up time with NST (n=21)) | 81 (the second group of 60 women was placed in the semi-Fowler position (Intervention 2) Allocated to intervention (n=81): Received allocated intervention (n=60) It was excluded because of insufficient follow-up time with NST (n=21)) | 143 (Since the women in this group were placed in the left lateral position that is routinely applied in the clinic in which the study was conducted, this was considered the control group. Allocated to intervention (n=143):Received allocated intervention (n=120) It was excluded because of insufficient follow-up time with NST (n=23))
Completed | 60 (Completion of electro monitoring application in the appropriate position) | 60 (Completion of electro monitoring application in the appropriate position) | 120 (Completion of electro monitoring application in the appropriate position)
Not Completed | 21 | 21 | 23
Not completed — Failure to complete the electro-monitoring application in the appropriate position | 21 | 21 | 23

BASELINE CHARACTERISTICS:
Population: The intervention group, comprising 120 pregnant women, was further divided into two subgroups: 60 women were assigned to the right lateral position, and 60 women to the semi-Fowler position. The control group, also consisting of 120 women, adhered to the clinic's routine practice of the left lateral position. All women in this group were placed in the left lateral position, with the remainder of the procedure conducted in the same manner as for the intervention groups.
Groups:
- Right Lateral Side-Lying Position; Semi-Fowler Position; Left Lateral Side-Lying Position: electro fetal monitoring
  Right side lying position: In the study, 60 participants were placed in the right side lying position (intervention 1)
  Semi Fowler: In the study, 60 participants in the semi-sitting position (intervention 2)
  left side lying position: In the study, 120 participants in the left side lying position (control group).
- Total: Total of all reporting groups
Arm/Group | Right Lateral Side-Lying Position | Semi-Fowler Position | Left Lateral Side-Lying Position | Total
Number analyzed (Participants) | 60 | 60 | 120 | 240
Age, Categorical [Count of Participants; unit: Participants]
  Age: <=18 years | 0 | 0 | 2 | 2
  Age: Between 18 and 65 years | 60 | 60 | 118 | 238
  Age: >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Geometric Mean (Standard Deviation); unit: years] | 31.62 (4.43) | 29.57 (3.93) | 30.24 (4.64) | 31.62 (4.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 120 | 240
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 60 | 60 | 120 | 240
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 60 | 60 | 120 | 240
Body Mass Index [Count of Participants; unit: Participants] — Body mass indexes of pregnant women were calculated.
  Participants
    30 and over (obese) | 12 | 12 | 28 | 52
    25-29 (overweight) | 32 | 28 | 61 | 121
    19-24 (normal) | 16 | 20 | 31 | 67
    18 and below (underweight) | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Right Side Lying Post NST (3)
Description: Blood Pressure (Systolic)-Blood pressure measurements were made before, during and after fetal monitoring of the pregnant women.
Time Frame: before NST
Measure: Geometric Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention 1 | Intervention 2 | Control Group
Number analyzed (Participants) | 60 | 60 | 120
mmHg | 113.67 (10.06) | 108.16 (10.56) | 112.80 (11.21)

2. Secondary Outcome: Right Side Lying
Description: Blood Pressure (Systolic)
Time Frame: NST instant
Measure: Geometric Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention 1 | Intervention 2 | Control Group
Number analyzed (Participants) | 60 | 60 | 120
mmHg | 110.37 (9.41) | 107.00 (8.57) | 108.89 (11.00)

3. Other Pre Specified Outcome: Right Side Lying
Description: Blood Pressure (Systolic)
Time Frame: post NST (NST time:1 minute)
Measure: Geometric Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention 1 | Intervention 2 | Control Group
Number analyzed (Participants) | 60 | 60 | 120
mmHg | 115.91 (10.76) | 100.08 (8.15) | 113.56 (12.28)

ADVERSE EVENTS:
Time Frame: 6 months
Description: There was no risk for any pregnant woman in the study.There is no risk for pregnant women participating in the study.
Arm/Group | Intervention 1 | Intervention 2 | Control Group
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/120
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/120

LIMITATIONS AND CAVEATS:
In the limited number of similar studies in the literature, it has been the supine position that has been examined but this has not produced robust results. For this reason, differing from other studies, the present study sought to examine the effects of the right lateral position and BMI on maternal blood pressure and fetal health.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT05863156/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT05863156/SAP_001.pdf